CLINICAL TRIAL: NCT07022054
Title: iCare IC1000 Alignment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icare Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TA032-168
Record Dates: First submitted 2025-05-22; First posted 2025-06-15 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Measurement of IOP Values (Experimental)
  Interventions: Device: iCare IC1000 measurement

INTERVENTIONS:
Device: iCare IC1000 measurement — Measurement of intraocular pressure with iCare IC1000

SUMMARY:
The primary objective of this study is to evaluate the performance of the alignment feature of iCare IC1000 tonometer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years

Exclusion Criteria:

1. Subjects with only one functional eye
2. Central corneal scarring
3. Microphthalmos
4. Buphthalmos
5. Contact lens use during measurement or hard lenses 24h prior to measurement
6. Dry eyes (clinically significant)
7. Nystagmus
8. Keratoconus
9. Any other corneal or conjunctival pathology or infection relevant to this study
10. Coloboma or other pupil deformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Primary Objective | Through study completion, an average of 2 months
  Number of participants with successful intraocular pressure (IOP) measurements using the alignment feature of the iCare IC1000 tonometer during a single clinic visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Clear Vue Laser Eye Center, Lake Worth, Florida, United States

IPD SHARING:
Plan to Share IPD: No